CLINICAL TRIAL: NCT04690881
Title: Psychodrama as a New Intervention for Treating Fear of Childbirth: a Randomized Controlled Trial
Brief Title: The Effect of Psychodrama for Treating Fear of Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Fadime Bayrı Bingöl, Phd. RN. Assistant Professor, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09.2018.672
Record Dates: First submitted 2020-12-28; First posted 2020-12-31 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Fear of Childbirth
Keywords: Fear of childbirth; Pychodrama; Psychoeducation; Childbirth-antenatal education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychodrama group psychoteraphy (Experimental): Psychodrama is not just a training but also a treatment technique where an individual is offered a potential cure, as well as improvement and awareness for his or her ongoing relationships within the group. In psychodrama, the participant is given an opportunity to re-experience of earlier incidents for a second time so that the person could be free from the impacts of that earlier experience. All of this happens simultaneously with joy, tears, laughter, and depth of feeling.Prenatal psychodrama is held by psychodrama psychotherapists in individual and group therapy sessions. In these sessions the pregnant mother encounters herself, her baby, her partner, her mother, her fear of childbirth and the moment of birth; she may act as protagonist in some scenes and in this way she closes any unfinished business from the past and rehearses the future in a safe therapeutic environment. In this study, 90-minute psychodrama practice was conducted in addition to pregnancy training for 6 weeks.
  Interventions: Behavioral: Psychodrama group psychotherapy
- Childbirth-antenatal education (No Intervention): Childbirth is one of the most significant events in a parent's life and has the potential to be an exhilarating and fulfilling experience for some or a frightening anxiety provoking experience for others. Structured antenatal classes have developed worldwide as traditional methods of information sharing have declined and expectant parents look for strategies to prepare for childbirth. In this study, routine pregnancy training was conducted for 6 weeks.

INTERVENTIONS:
Behavioral: Psychodrama group psychotherapy — In order to reduce the fear of cihildbirth, pregnant women are given 90 minutes right after the training in addition to the routine pregnancy training. In the psychodrama-based pregnancy education program, fear of childbirth were assesment by sociometric measurement in order to increase the awareness of pregnant women about birth fear levels in the first week. Afterwards, they were given the opportunity to express themselves about the factors that may cause fear in pregnant women (their previous traumatic experiences, negative prejudices about childbirth, etc). The group members shared about their process in the first session and the session was ended. The session was evaluated with other researchers. In the following sessions, in order to strengthen their coping with the fear of childbirth, besides psychodrama warm-up games, the basic techniques of psychodrama, role switching, matching and mirror were used in protogonist works.
  Arms: Psychodrama group psychoteraphy

SUMMARY:
This study is a randomized controlled study. This research was carried out with the aim of determining the effect of psychodrama-based pregnancy education program on fear of childbirth (FOC). The population of the study consisted of 18-45 years old pregnant who with high fear of childbirth. The sample of the study was determined as 150 pregnant with confidence level of 95% and theoretical power of 95%. The pregnant women were divided into two groups of 75 pregnant. In addition to routine pregnancy training, a 90-minute psychodrama study was carried out to the experimental group. Data were collected using the information form, Wijma Delivery Expectancy/ Experience Questionnaire Version A (W-DEQ), Wijma Delivery Expectation / Experience Questionnaire Version B (W-DEQ), City Birth Trauma Scale and Edinburgh Postpartum Depression Scale. The data obtained were assesment using the SPSS (Version 21.0) package program on the computer.

DETAILED DESCRIPTION:
The pregnant women were divided into two groups of 75 pregnant. In addition to the 6-week routine pregnancy training, a 90-minute psychodrama study was conducted to the experimental group. The experimental group was divided into 6 subgroups and trained (min = 9, max = 14). The control group was divided into 6 subgroups and trained (min = 11, max = 14). Prenatal psychodrama is held by psychodrama psychotherapists in individual and group therapy sessions. In these sessions the pregnant mother encounters herself, her baby, her partner, her mother, her fear of childbirth and the moment of birth; she may act as protagonist in some scenes and in this way she closes any unfinished business from the past and rehearses the future in a safe therapeutic environment.Data were collected using the information form, Wijma Delivery Expectancy/ Experience Questionnaire Version A (W-DEQ), Wijma Delivery Expectation / Experience Questionnaire Version B (W-DEQ), City Birth Trauma Scale and Edinburgh Postpartum Depression Scale. The data obtained were assesment using the SPSS (Version 21.0) package program on the computer.

ELIGIBILITY:
Inclusion Criteria:

* willing to participate in the study voluntarily,
* non-disabled (hearing, seeing, understanding),
* having 38 or more points from Wijma Birth Experience / Expectation Scale A,
* living with his wife,
* primipary,
* not diagnosed with risky pregnancy and
* women with suitable weeks of gestation (between 20-30 weeks) were included in the study.

Exclusion Criteria:

* those who were diagnosed with risky pregnancy during the training,
* did not attend the first week of the pregnancy training program,
* were absent for more than a week,
* had difficulty following group studies,
* completed the forms incompletely, and
* did not want to continue working / gave up from the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant
Enrollment: 150 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Fear of childbirth | 6 week
  Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ): The minimum and maximum scores that can be obtained from the questionnaire are 0 and 165, respectively. Higher scores indicate greater levels of Fear of Childbirth.
Fear of Childbirth | Postpartum 7-14 days
  Wijma Delivery Expectancy/Experience Questionnaire version B: The minimum and maximum scores that can be obtained from the questionnaire are 0 and 160, respectively. Higher scores indicate greater levels of Fear of Childbirth.

SECONDARY OUTCOMES:
Postpartum posttraumatic stress | Postpartum 6. Months
  City Birth Trauma Scale:Total scores can range from 0 to 60. Higher scores are indicative of a greater number of Post Traumatic Stress Disorder symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Fadime Bingöl, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No